CLINICAL TRIAL: NCT07100171
Title: A Single-Center, Open-Label, Single-Arm Exploratory Study Evaluating GM101 Injection in Patients With Mid-to-Late Stage Parkinson's Disease
Brief Title: Evaluation of GM101 Injection in Patients With Parkinson's Disease
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Genemagic Biosciences Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202411203-4
Record Dates: First submitted 2025-02-18; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Parkinson's Disease

STUDY DESIGN:
Intervention Model Description: This is a dose-escalation study with two dose cohorts under a single-group assignment framework
Masking Description: Masking Description
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental: GM101 dose escalation (Experimental): This is a dose-escalation study with two dose cohorts under a single-group assignment framework
  Interventions: Other: Biological: GM101

INTERVENTIONS:
Other: Biological: GM101 — Neurosurgical delivery of GM101 to the putamen

SUMMARY:
The objective of this study is to assess the safety of GM101 in participants with Parkinson's disease (PD)

DETAILED DESCRIPTION:
We utilize adeno-associated viruses (AAVs) to deliver gene to reprogram astrocytes in the putamen into dopaminergic neurons to treat patients with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

1. Clinically diagnosed patients with primary Parkinson's Disease [in accordance with the "Diagnostic Criteria for Parkinson's Disease in China" released in 2016];
2. Participants must be able to comprehend (fully understand the details of the clinical trial and the potential risks and benefits of the study) and voluntarily sign the informed consent form. When participants are unable to read, the informed consent form and other written materials may be read by a legal representative or an impartial witness, who will also witness the consent process;
3. Age between 40 and 70 years old, inclusive, regardless of gender;
4. Body weight between 40 kg and 110 kg, and Body Mass Index (BMI) between 18 kg/m² and 34 kg/m²;
5. A history of Parkinson's Disease for >= 5 years;
6. Able to undergo surgical anesthesia, suitable for neurosurgical procedures under anesthesia, and capable of undergoing CT/MRI examinations;
7. Hoehn-Yahr stage (Appendix IV Hoehn-Yahr Staging) at screening in the "off" state is 4-5 (including borderline values);
8. MDS-Unified Parkinson's Disease Rating Scale Part III Motor Examination (MDS-UPDRS-III) score in the "off" state >= 30; and a positive levodopa challenge test (improvement in UPDRS-III score from "off" to "on" state >30%);
9. Patients whose PD symptoms cannot be effectively controlled or who experience intolerable adverse drug reactions despite treatment with medications recommended by the "Chinese Guidelines for the Treatment of Parkinson's Disease (4th Edition)-2020";
10. Receiving a stable dose of anti-Parkinson's medication for at least 4 weeks prior to administration;
11. Acceptable laboratory values during the screening period and prior to administration (Day 0): a) Hemoglobin >= 100 g/L; b) Platelets >= 100×10^9/L; c) Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) <= 1.5 times the upper limit of normal; d) Total bilirubin <= 1.5 times the upper limit of normal; e) Serum creatinine (Cr) <= 1.5 times the upper limit of normal;
12. Participants agree not to receive any other therapeutic intervention studies during the main study phase;
13. Participants agree not to participate in any other clinical studies during the study period;
14. Participants agree not to receive any other vaccines within 30 days after administration;
15. Participants must have the ability to live independently or the ability to clearly delegate relevant caregivers, with good compliance, and be able to attend regular follow-ups. During follow-up, participants must accurately complete the PD patient diary, and family members, guardians, or caregivers may assist in filling out the patient diary;
16. Participants must have a pre-existing neutralizing AAV8 antibody titer <= 1:90 as determined by testing;
17. Based on the judgment of the Principal Investigator (PI), cancer-related screening will be conducted for patients who meet the inclusion criteria.

Exclusion Criteria:

1. Patients with atypical parkinsonian syndromes (Parkinson-plus syndromes, secondary Parkinson's syndrome, or hereditary Parkinson's syndrome).
2. Patients who have previously undergone pallidotomy, deep brain stimulation (DBS) surgery, striatal/extrapyramidal system surgery, stereotactic brain surgery, or other cerebral surgeries that might affect the observation of this trial's outcomes; or those who have undergone other surgeries deemed by investigators to interfere with study participation.
3. Patients with intracranial lesions revealed by previous CT/MRI scans, such as cerebral trauma, cerebrovascular malformations, hydrocephalus, brain tumors, or striatal/other brain region abnormalities that significantly increase surgical risks.
4. Patients with history of the following cardiovascular/cerebrovascular diseases: 1)Severe heart failure, unstable angina, or myocardial infarction; 2)Severe arrhythmias including but not limited to II/III-degree atrioventricular block or prolonged QT interval; 3)Long QT syndrome; 4)Cardiovascular surgery history; 5)History of stroke or transient ischemic attack (TIA) within 3 months, deemed ineligible by investigators; 6)Subarachnoid hemorrhage history; 7)Major vascular diseases considered ineligible by investigators.
5. Patients with history of malignant tumors.
6. Patients who have received cell therapy.
7. Patients who have received gene therapy.
8. Patients with active disseminated intravascular coagulation or significant bleeding tendency within 3 months prior to consent, or those unable to discontinue antiplatelet/anticoagulant medications >= 7 days pre-operation, or whose coagulation function hasn't normalized >= 10 days after stopping antiplatelet medications.
9. Patients who received prolonged >= 14 days) high-dose systemic corticosteroids (prednisone >= 20 mg/day or equivalent) or immunosuppressants within 3 months prior to consent (topical use excluded).

10,Patients with psychiatric disorders deemed ineligible by investigators; or those with suicidal ideation/attempts (including actual attempts, interrupted attempts, or aborted attempts) within the past year or currently.

11.Patients who received botulinum toxin treatment within 6 months prior to consent.

12.Patients with active epilepsy or currently using antiepileptic drugs. 13.Patients with dementia or severe cognitive impairment history; or those showing significant dementia/cognitive dysfunction during screening; MDS-UPDRS Part 1.1 cognitive impairment score >3; dementia affecting compliance, diary accuracy, and/or informed consent capability.

14. Individuals with severe depression (Hamilton Depression Rating Scale [HAM-D17] score >= 24) or severe anxiety (Hamilton Anxiety Rating Scale [HAMA] score >= 29) during screening.

15. Individuals with the following clinically significant abnormalities during screening: 1) Abnormal coagulation function (prothrombin time >= 1.5 times the upper limit of normal, activated partial thromboplastin time >= 1.5 times the upper limit of normal); 2) Clinically significant immunological abnormalities, deemed unsuitable for participation by the investigator; 3) Poorly controlled hypertension (defined as blood pressure remaining above 160/100 mm Hg despite antihypertensive treatment) and severe orthostatic hypotension; 4) Poorly controlled diabetes (glycated hemoglobin > 9.0%, or fasting plasma glucose [FPG] >= 11.1 mmol/L).

16. Individuals with surgical contraindications (e.g., prior cochlear implant, pacemaker, defibrillator, stereotactic neurosurgery, or prior implantation of unilateral or bilateral similar devices) or those who have undergone other surgeries within the past six months that the investigator believes may affect the trial, or those with allergies (e.g., to contrast agents) preventing MRI, or other neurosurgical contraindications.

17. Individuals with other severe systemic diseases, such as cor pulmonale, severe chronic obstructive pulmonary disease (COPD) (FEV1% < 50%), etc.

18. Individuals with any of the following conditions: positive human immunodeficiency virus (HIV) antibody; positive syphilis antibody; positive hepatitis C virus (HCV) antibody with detectable HCV RNA; positive hepatitis B virus surface antigen with HBV DNA copy number above the normal limit; active tuberculosis; or other active infections deemed by the investigator to potentially affect participation or study outcomes.

19. Individuals with alcohol addiction, positive drug abuse screening, or a history of drug dependence.

20. Individuals with contraindications or allergies to any components of the drugs used in the study (e.g., tacrolimus, levodopa) or to similar drugs or other macrolide drugs, or those with a history of allergies (e.g., to two or more drugs or foods).

21. Women of childbearing potential or breastfeeding women who have not undergone sterilization, are not postmenopausal, or are unwilling to use medically approved effective contraception for two years after receiving the study drug, and men who have not undergone sterilization or are unwilling to use medically approved effective contraception for two years after receiving the study drug.

22. Individuals who have received electroconvulsive therapy within 30 days prior to dosing.

23. Individuals currently participating in other clinical trials or those who have participated in other clinical studies and received interventional treatment within three months prior to dosing.

24. Individuals deemed by the investigator to have poor compliance. 25. Patients currently receiving treatment such as apomorphine or levodopa infusion therapy (Duodopa®).

26. Individuals with severe movement disorders in both medicated and unmedicated states.

27. Individuals with major illnesses or any other conditions deemed by the investigator to jeopardize the safety of the participant or affect the investigator's assessments.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-05-29 (Actual); Primary Completion 2027-02-17 (Estimated); Study Completion 2030-02-17 (Estimated)

PRIMARY OUTCOMES:
Grading of adverse Events/Serious Adverse Events (AE's/SAE's) | Baseline to 5 Years After Gene Transfer
  Grading will be assessed using NCI CTCAE, version 4.03. Grade 1 = Mild Grade 2 = Moderate Grade 3 = Severe Grade 4 = Potentially life-threatening Grade 5 = Death

SECONDARY OUTCOMES:
Change in motor function using Unified Parkinson's Disease Rating Scale (UPDRS); | Baseline to 5 Years After Gene Transfer
  Standard assessment scale used to quantify signs and symptoms of PD. The total UPDRS score is calculated by summing the scores from each section, ranging from 0 (no disability) to 176 (severe disability), the higher scores indicate the greater severity of symptoms.
Change in motor function using Modified Hoehn and Yahr Scale | Baseline to 5 Years After Gene Transfer
  Scale used to measure overall level of disability due to PD. The scale includes stages 1 through 5, the higher stage means the worse condition.
Change in occurrence of dyskinesia using Unified Dyskinesia Rating Scale (UDysRS) | Baseline to 5 Years After Gene Transfer
  Comprehensive rating tool used to assess essential features of dyskinesia in PD.
Change in Parkinson's medications | Baseline to 5 Years After Gene Transfer
  Change in Parkinson's medications compared to Baseline.
Change in dopamine transporter binding assessed by regional brain using [¹¹C]CFT-PET (DAT imaging) | Baseline to 5 Years After Gene Transfer
  Change in Parkinson's DAT imaging compared to Baseline.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital, Central South University, Changsha, China

IPD SHARING:
Plan to Share IPD: No